CLINICAL TRIAL: NCT00801255
Title: A Randomized, Placebo-controlled, Dose-ranging Study to Evaluate the Safety, Tolerability and Antiviral Activity of Combination Treatment With an HCV Polymerase Inhibitor (RO5024048) and an HCV Protease Inhibitor (RO5190591) in Genotype 1 Chronic Hepatitis C Patients. INFORM 1
Brief Title: A Study of Combination Treatment With an HCV Polymerase Inhibitor (RO5024048) and an HCV Protease Inhibitor (RO5190591/Danoprevir) in Genotype 1 Chronic Hepatitis C Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PP22205
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — danoprevir

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (7):
- Cohort A (Experimental)
  Interventions: Drug: RO5024048
- Cohort B (Experimental)
  Interventions: Drug: danoprevir
- Cohort C (Experimental)
  Interventions: Drug: danoprevir
- Cohort D (Experimental)
  Interventions: Drug: danoprevir
- Cohort E (Experimental)
  Interventions: Drug: danoprevir
- Cohort F (Experimental)
  Interventions: Drug: danoprevir
- Cohort G (Experimental)
  Interventions: Drug: danoprevir

INTERVENTIONS:
Drug: RO5024048 — 500mg po bid/100mg po q8h for 7 days
  Arms: Cohort A
Drug: danoprevir — 500mg po bid/100mg po q8h for 14 days
  Arms: Cohort B
Drug: danoprevir — 1000mg po bid/100mg po q8h for 14 days\n500mg po bid/200mg po q8h for 14 days
  Arms: Cohort C
Drug: danoprevir — 1000mg po bid/200mg po q8h for 14 days
  Arms: Cohort D
Drug: danoprevir — 1000mg/600mg po twice daily for 14 days
  Arms: Cohort E
Drug: danoprevir — 1000mg/900mg po twice daily for 14 days
  Arms: Cohort F; Cohort G

SUMMARY:
This 7 cohort study will evaluate the efficacy and safety of combination treatment with an HCV nucleoside polymerase inhibitor(RO5024048)and an HCV protease inhibitor(RO5190591/ITMN-191/danoprevir) in patients with chronic hepatitis C, genotype 1.Cohorts A,B,C,D and G will be treatment-naive patients, cohort E will be treatment-experienced excluding null responders, and cohort F will be null responders. Cohorts A and B will evaluate doses of 500mg po bid RO5024048 and 100mg po q8h RO5190591, alone or in combination, for up to 7 or 14 days. Cohort C will evaluate combination treatment with either 1000mg po bid RO5024048 and 100mg q8h RO5190591 or 500mg po bid RO5024048 and 200mg q8h RO5190591 for 14 days. Cohort D will evaluate 1000mg po bid RO5024048 and 200mg q8h RO5190591 for 14 days.Cohort E will evaluate 1000mg RO5024048/600mg RO5190591 po twice daily for 14 days, and Cohorts F and G will evaluate 1000mg RO5024048/900mg RO5190591 po twice daily for 14 days. Cohorts will be tested sequentially or in parallel, if supported by appropriate safety and pharmacokinetic data.Following the last dose of study medication patients have the option of continuing treatment with Standard of care therapies. The anticipated time on study treatment is <3 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-65 years of age;
* chronic hepatitis C, genotype 1.

Exclusion Criteria:

* decompensated liver disease, or impaired liver function;
* presence or history of non-hepatitis C chronic liver disease;
* HBsAg or HIV infection;
* history of cancer within 5 years, other than localized or in situ cancer of the skin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2008-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
HCV RNA | At each clinic visit, throughout study
Adverse events, laboratory parameters, vital signs | At each clinic visit, throughout study

SECONDARY OUTCOMES:
PK parameters;viral resistance | At intervals, throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Australia (3):
  - Adelaide
  - Heidelberg
  - Melbourne
- New Zealand (2):
  - Christchurch
  - Grafton

REFERENCES:
- [Derived] Gane EJ, Roberts SK, Stedman CA, Angus PW, Ritchie B, Elston R, Ipe D, Morcos PN, Baher L, Najera I, Chu T, Lopatin U, Berrey MM, Bradford W, Laughlin M, Shulman NS, Smith PF. Oral combination therapy with a nucleoside polymerase inhibitor (RG7128) and danoprevir for chronic hepatitis C genotype 1 infection (INFORM-1): a randomised, double-blind, placebo-controlled, dose-escalation trial. Lancet. 2010 Oct 30;376(9751):1467-75. doi: 10.1016/S0140-6736(10)61384-0. Epub 2010 Oct 14. PMID 20951424